CLINICAL TRIAL: NCT03491189
Title: Helical Blade vs Lag Screw Fixation for Intertrochanteric Hip Fractures: A Prospective Randomized Controlled Study
Brief Title: Blade vs Screw Intertrochanteric Hip Fracture Fixation Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol change
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Garner, Assistant Professor, Department of Orthopaedics, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00008033
Record Dates: First submitted 2018-03-29; First posted 2018-04-09 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Pertrochanteric Fracture of Femur, Closed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lag screw fixation (Active Comparator): Lag screw fixation
  Interventions: Device: Lag screw fixation
- Helical Blade fixation (Active Comparator): Helical Blade fixation
  Interventions: Device: Helical blade fixation

INTERVENTIONS:
Device: Lag screw fixation — surgical fixation
  Other Names: Cephalomedullary Hip Screw
  Arms: Lag screw fixation
Device: Helical blade fixation — surgical fixation
  Other Names: Cephalomedullary Blade
  Arms: Helical Blade fixation

SUMMARY:
This study evaluates the rate of cut-out and fixation failures in helical blade fixation versus lag screw fixation for cephalomedullary nailing of peritrochanteric femur fractures.

DETAILED DESCRIPTION:
As the population ages, the prevalence of peritrochanteric femur fractures continues to increase each year. An increase in the use of intramedullary devices as treatment has accompanied this increase in peritrochanteric femur fractures. Intramedullary devices are now used more frequently than plate and screw constructs nationwide to treat peritrochanteric femur fractures1. While the prognosis following intramedullary device placement remains favorable compared to other treatment options, there are still complications that exist. Cut-out of the cephalomedullary implant through the femoral head has long been one of the more prevalent complications when using an intramedullary device.2 To address the shortcomings that cause lag screw cut-out, the helical blade was designed. In theory, it provides improved fixation over the lag screw by compacting cancellous bone as it is inserted and may also be more effective at supporting torsional loading.3 Additionally, the helical blade has been shown to require less operation time and less fluoroscopy time during implantation.4

Currently, there is a lack of a randomized prospective study comparing the rates of cut-out in lag screw fixation and helical blade fixation of peritrochanteric femur fractures using third generation cephalomedullary femoral nails. A recent retrospective study by Stern et al analyzed the rate of cut-out of helical blades and lag screws in peritrochanteric femur fractures treated with cephalomedullary nails and found that the helical blade was much more prone to cut-out than the lag screw. Cut-out rates were 15.1% and 3.0% for the implants respectively.5 While this study seems to suggest that, in terms of cutout, the helical blade is inferior to the lag screw, there are many factors that limit its validity and applicability. First, the study was a retrospective study which inherently induces some level of bias. Next, the study recorded a cut-out rate for the helical blade that is much higher than and not consistent with studies that have been previously reported. Flores et al reported a cut-out rate of 3.4% in 258 patients treated with the helical blade, Gardner et al reported a cut-out rate of 5.15% in 97 patients treated with the helical blade, and Liu et al reported a cut-out rate of 6.7% in 223 patients treated with the helical blade.6,7,8 These numbers are all drastically lower than the rates of cut-out reported by Stern et al. Another limitation to their study was that 26 surgeons operated on the 362 patients that were included in the study. This large number of surgeons introduced a significant amount of variability that could not be controlled for. While this study provides some evidence that the helical blade may be inferior to the lag screw in terms of cut-out, it is not definitive and a prospective study is needed to truly validate this claim. Additionally, factors such as tip-apex distance, time to cut-out, direction of cut-out reduction quality, and fracture pattern must be analyzed to accurately assess the usefulness of the helical blade compared to the lag screw and determine predictors for cut-out.

While the primary purpose of this study will be to analyze rates of cut-out between the two fixation devices, we are also interested in determining a threshold tip-apex distance that is predictive of cut-out. While Stern et al reported data that supported the hypothesis that increased tip-apex distance is predictive of cut-out, they did not identify a threshold that, itself, is predictive of cut-out.5 It was previously thought that a tip-apex distance greater than 25mm is predictive of cut-out.4 Other studies, however, have shown that tip-apex distances that are too small are also predictive of cutout.8 It will be our goal to measure tip-apex distance in all patients and attempt to determine if there is a threshold that is predictive of cut-out.

Another factor of importance that we will investigate is the direction of cut-out of the two implants. Previous comparisons have found that while the lag screw tends to cutout superiorly, the helical blade is much more likely to cutout medially.5,8 This is thought to be due to the compaction of bone that occurs when the helical blade is inserted and also why there appears to be greater rates of cut-out with smaller tip-apex distances.8 By gaining a further understanding of the direction that these implants typically fail we hope to have another predictor of cut-out.

Finally, it will be our goal to attempt to assess reduction quality and fracture pattern to determine each factor's predictive value of cut-out. It has already been suggested that non-anatomical reduction and complex fracture patterns increase the likelihood of cut-out.9

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with low-energy peritrochanteric femur fractures
* Age 55 years and older
* Sex: male or female

Exclusion Criteria:

* Non English speaking
* Age < 55 years

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2018-06-19 (Actual); Study Completion 2018-06-19 (Actual)

PRIMARY OUTCOMES:
Implant cut-out | 12 months
  Rate of implant cut-out after cephalomedullary nailing of peritrochanteric femur fractures in a randomized prospective study.

IPD SHARING:
Plan to Share IPD: No